CLINICAL TRIAL: NCT03535142
Title: Prognostic Significance of Fatty Liver Disease in Bariatric Patients
Acronym: PROMETHEUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other); Esbjerg University Hospital of South-West Jutland (Unknown)
Responsible Party: Principal Investigator, Mette Munk Lauridsen, Associate professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20170210
Record Dates: First submitted 2018-05-01; First posted 2018-05-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Metabolic Encephalopathy; Obesity, Morbid; Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Brain Diseases, Metabolic; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention is bariatric surgery (Roux en Y gastric bypass or gastric sleeve operation).
  Interventions: Procedure: Bariatric surgery
- Control (No Intervention): Age, BMI and co-morbidity matched group who do not undergo surgery.

INTERVENTIONS:
Procedure: Bariatric surgery — Roux en y gastric bypass or gastric sleeve operation
  Arms: Intervention

SUMMARY:
Prospective non-randomized intervention case control study on patients with a BMI > 35. The intervention group/cases (n=600) is comprised of bariatric patients who undergo bariatric surgery and the control group (n=600) of age, weight and comorbidity matched patients who choose not to undergo bariatric surgery. The overall aim is to examine prevalence of the spectrum of fatty liver disease (NAFLD) in these patients and the prognostic significance of NAFLD.

ELIGIBILITY:
Inclusion Criteria case group:

* Age > 18 years
* BMI >35 kg/m2 and referred for bariatric surgery at Hospital of South West Jutland, Denmark
* Able to give written informed consent.

Inclusion criteria control group:

* Age > 18 years
* BMI >35 kg/m2 with no wish to undergo bariatric surgery.
* Able to give written informed consent.

Exclusion Criteria:

* Active viral hepatitis
* Not willing or able to consent
* Contraindications to liver biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2035-06-01 (Estimated); Study Completion 2038-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will die during the follow up period in case and control group | 10 years follow up after inclusion
  Difference in mortality between cases and controls with various NAFLD severity on biopsy.

SECONDARY OUTCOMES:
Number of participant who will experience progressive fatty liver disease in case and control group | 10 years follow up after inclusion
  Difference NAFLD severity between case and control group after 10 years follow up. Simple steatosis is the mildest form and liver cirrhosis is the most serious manifestation:
  1. Grade 1 steatosis
  2. Grade 2 steatosis
  3. Grade 3 steatosis
  4. Non alcoholic steatohepatitis
  5. Presence of fibrosis Kleiner grade 1-2
  6. Presence of fibrosis Kleiner grade 3
  7. Presence of liver cirrhosis
Change in continuous reaction time measurement after bariatric surgery | 10 years follow up after inclusion
  Continuous reaction time measurement will measure reaction time instability and is a measure of metabolic encephalopathy. The method is a 10-minutes, computerised registration of a series of motor reaction times to an auditory stimulus, with results reported as the CRTindex (50 percentile/(90-10) percentile) as a parameter of reaction time variability. A CRT index below 1.9 i considerede abnormal a may be a sign of hepatic encephalopathy.
Change in EEG after bariatric surgery | 24 months after surgery
  Change in mean dominant frequency(MD) on EEG spectral analysis. EEG disturbances in hepatic encephalopathy are (rated by severity)but there is no enough space here to describe it.
Change in intelligence quotient after bariatric surgery | 24 months efter surgery
  Measured by Weschlers adult intelligence scale (WAIS). An IQ if 100 i the norm. Range 50-150.

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Lauridsen, MD, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of Southwest Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wernberg CW, Indira Chandran V, Lauridsen MM, Skytthe MK, Hansen CD, Hansen JK, Gronkjaer LL, Jacobsen BG, Di Caterino T, Detlefsen S, Thiele M, Guiliani AM, Villesen IF, Leeming DJ, Karsdal M, Graversen JH, Krag A. Ability of soluble TREM2 and PRO-C3 as biomarkers to predict changes in MASLD activity. JHEP Rep. 2025 Apr 22;7(8):101432. doi: 10.1016/j.jhepr.2025.101432. eCollection 2025 Aug. PMID 40677693